CLINICAL TRIAL: NCT02786524
Title: A Randomized Study to Evaluate the Effect of Outpatient Symptom Management on Symptom Burden in Advanced Stage or Recurrent Gynecologic Oncology Patients Receiving Chemotherapy
Brief Title: Effect of Outpatient Symptom Management on Gynecologic Oncology Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Katherine Harris, Gynecologic Oncology Fellow, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00089412
Record Dates: First submitted 2016-05-10; First posted 2016-06-01 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Uterine Cervical Neoplasms; Ovarian Neoplasms; Gynecologic Neoplasms; Fallopian Tube Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Peritoneal Neoplasms
Keywords: Palliative Care; Triage; Symptom Evaluation; Chemotherapy; Patient Distress
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Genital Neoplasms, Female; Fallopian Tube Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Peritoneal Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): Patients randomized to this arm receive standard symptom management care by their primary gynecologic oncologist and complete the NCCN distress thermometer and ESAS-r at each visit, every 3-4 weeks.
- Symptom Management and Supportive Care (Experimental): Patients randomized to this arm are referred to a specialized symptom management and supportive care clinic and seen within two weeks. Patients will be seen in follow-up as recommended by the symptom management providers, and at each visit they will complete the ESAS-r and NCCN distress thermometer and return their responses either in person or by mail to the study team in a pre-addressed postage paid envelope.
  Interventions: Behavioral: Specialized Symptom Management and Supportive Care

INTERVENTIONS:
Behavioral: Specialized Symptom Management and Supportive Care — Based on Patients who score 5 or higher on the Baseline Patient Palliative Care Survey that will identify patients that will most benefit from specialty palliative care
  Arms: Symptom Management and Supportive Care

SUMMARY:
To evaluate whether formal referral to The Symptom Management and Supportive Care Clinic improves symptom burden in advanced stage or recurrent gynecologic oncology chemotherapy patients compared with symptom management performed by the primary gynecologic oncologist.

DETAILED DESCRIPTION:
Patients with gynecologic malignancies often have a high prevalence of symptoms throughout their disease course including fatigue, pain, anxiety and depression. Palliative care is defined by the World Health Organization (WHO) as "an approach that improves the quality of life of patients and their families facing the problems associated with life threatening illness, through the prevention and relief of suffering by means of early identification and impeccable assessment and treatment of pain and other problems, physical, psychosocial and spiritual."

The University of Michigan Symptom Management and Supportive Care Program works together with patient's oncology team to manage cancer related and treatment related symptoms. They offer a wide range of services including: pain and symptom management, medication management, nutritional counseling, expedited access to psychiatric oncology, anesthesia pain service and physical medicine and rehabilitation. Studies have demonstrated an improvement in quality of life, symptom burden and patient/care giver satisfaction when palliative care is part of routine oncologic care. Currently, in gynecologic oncology, palliative care is incorporated on a case by case basis, instead of in a standardized approach. We hope this study will provide a standardized tool to identify gynecologic oncology patients receiving chemotherapy who would benefit from a referral to a symptom management clinic.

This study will provide a screening mechanism to identify advanced stage or recurrent gynecologic oncology chemotherapy patients with palliative care needs and determine which symptom management option provides the best improvement in symptom burden, that performed by a specialty clinic staffed by providers formally trained in palliative care or that provided by the patient's gynecologic oncologist. This study has the potential to change practice by providing a triage tool that will identify patients that will most benefit from specialty palliative care services and could result in improved quality of life for our patients.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Diagnosis of Stage III, IV, or recurrent gynecologic malignancy (Uterine, Ovarian, Cervical, Vulvar, Vaginal, Fallopian Tube, Primary Peritoneal)
* Receiving active intravenous, intraperitoneal, or oral chemotherapy
* Patient at University of Michigan Gynecologic Oncology Clinic

Exclusion Criteria:

* Male
* Less than 18 years of age
* Patients without a diagnosis of a gynecologic malignancy
* Patients not receiving intravenous, intraperitoneal or oral chemotherapy at the time of enrollment
* Patients receiving radiation therapy with chemo-sensitization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Symptom Burden as Determined by the Edmonton Symptom Assessment System | Baseline and 3 months after study start
  To determine if referral to a symptom management clinic improves the symptom burden quantified by the patients' Edmonton Symptom Assessment System (ESAS) scores.
Change in Patient-Reported Symptom Burden as Determined by the National Comprehensive Cancer Network Distress Screening Tool | Baseline and 3 months after study start
  To determine if referral to a symptom management clinic improves the symptom burden quantified by the patients' National Comprehensive Cancer Network (NCCN) Distress Screening Tool scores.

SECONDARY OUTCOMES:
Baseline Symptom Burden and Palliative Care Needs | Baseline
  To determine the baseline symptom burden and palliative care needs upon enrollment of patients with advanced stage or recurrent gynecologic malignancies receiving chemotherapy.
Change in Patient-Reported Distress | 3 months after study start, 6 months after study start, and 9 months after study start
  Measure changes in patient-reported distress using the NCCN Distress Thermometer
Change in Symptom Burden | 6 months after study start and 9 months after study start
  Evaluate changes in patients' symptom burden with the ESAS-r to evaluate the ongoing sustained effect of the intervention.
Change in Patient Adherence to Symptom Management Program | 6 months after study start and 9 months after study start
  To analyze patients in the symptom management arms with a 3-item questionnaire to determine what factors are associated with adherence to a symptom management program.
Barriers to Symptom Management and Supportive Care | 9 months after study start
  Analyze barriers that prevented patients from attending the Symptom Management and Supportive Care Clinic, as identified in a 3-item questionnaire.
Overall Survival Rate | Upon study completion, an average of 1 year
  Overall survival will be compared between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Harris, MD, Principal Investigator — University of Michigan; Carolyn M Johnston, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No